CLINICAL TRIAL: NCT03915938
Title: Ketamine's Effect Changes the Cortical Electrophysiological Activity Related to Semantic Affective Dimension of Pain: a Placebo-controlled Study in Healthy Male Subjects
Brief Title: Ketamine's Effect Changes the Cortical Electrophysiological Activity Related to Semantic Affective Dimension of Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-0019
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2018-01

CONDITIONS: Acute Pain; Chronic Pain, Widespread; Schizophrenia
Keywords: Ketamine; ERP; Oddball
MeSH Terms: conditions — Acute Pain; Chronic Pain; Schizophrenia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group S-Ketamine (Experimental): S-Ketamine will be diluted in normal saline and administrated in a target controlled infusion using an infusion pump to obtain a plasma target of 60 ng/ml according to Domino's model. Infusion will start during the interval between the 3rd and 4th blocks of the task.
  Interventions: Drug: Ketamine
- Group Placebo (Placebo Comparator): A previously prepared identical solution containing only normal saline will be infused at the same infusion rates of group ketamine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — S-ketamine will be administered in precalculated infusion rates to obtain a plasmatic level of 60 ng/ml
  Arms: Group S-Ketamine
Drug: Placebo — Administered in an identical way than ketamine.
  Arms: Group Placebo

SUMMARY:
This is a clinical trial that intend to determine the effects of S-ketamine on event-related potentials associated with semantic affective pain-processing

DETAILED DESCRIPTION:
Ketamine is a unique anesthetic with neural effects that are distinct from more commonly-used γ-aminobutyric acid agonists. Evidence suggest that analgesic effect of ketamine is primarily related to the affective than the sensorial aspects of pain interpretation. The investigators investigated whether ketamine, a noncompetitive NMDA antagonist, would modify the perceived emotional valence of pain-related words when compared to non-pain-related ones in healthy volunteers. Using a single session double-blind parallel placebo-controlled design, 24 healthy volunteers were randomized to receive intravenous S-ketamine (n=12) or placebo (n=12). During infusion (plasmatic target of 60 ng/ml), the effects of ketamine were recorded using EEG and oddball behavioral data was monitored. Evoked potentials (N200 and P300 components) were recorded during performance of a semantic written word oddball task containing pain-related (targets) and non-pain-related words (standards). Expected results: The findings of this study can help in the understanding of neurophysiologic mechanisms involved in ketamine's effects both in psychiatric diseases as in the treatment of postoperative acute and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* male healthy subjects with higher education level

Exclusion Criteria:

* do not understand Portuguese language
* obese patients (BMI > 27 kg/m2)
* use of NSAID, steroids, analgesics, anticonvulsant drugs, as well as alpha and beta-blockers
* score ≥ 13 on Beck II Questionnaire
* sleep deprivation in the night before evaluation

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
AUC of the grand averaged mean differences between ERPs elicited by target and non-target words | up to 60 min
  EEG will be recorded during all task time. The main outcome will be the area under de curve (AUC) of the grand averaged mean differences between event-related potencials (ERPs) elicited by target and non-target words at 100-200, 300-500 and 800-900 ms after stimulus presentation for parietal electrophysiological signal (Pz). The ERPs represent the averaged voltage of several trials.

SECONDARY OUTCOMES:
Word ratings related to the semantic valence | up to 60 min
  After viewing each word, volunteers were asked to classify them according to the semantic valence in the following categories: "positive," "negative" or "neutral."
Response times (behavioural oddball data) | up to 60 min
  Response times to word classification in oddball task

OTHER OUTCOMES:
Subjective euphoria rating | up to 60 min
  Euphoria will be rated using an analogue visual scale ranging of 0 to 10.
Subjective sedation rating | up to 60 min
  Sedation will be rated using an analogue visual scale ranging of 0 (completely awake) to 100 (sleeping).

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schwertner A, Zortea M, Torres FV, Ramalho L, Alves CFDS, Lannig G, Torres ILS, Fregni F, Gauer G, Caumo W. S-Ketamine's Effect Changes the Cortical Electrophysiological Activity Related to Semantic Affective Dimension of Pain: A Placebo- Controlled Study in Healthy Male Individuals. Front Neurosci. 2019 Sep 13;13:959. doi: 10.3389/fnins.2019.00959. eCollection 2019. PMID 31611759